CLINICAL TRIAL: NCT03592160
Title: Role of Rehabilitation for the Repair of Pelvic Floor Injuries Associated to Vaginal Delivery Identified by 3/4D Transperineal Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Valme (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, José Antonio García Mejido, Principal Investigator, Hospital Universitario de Valme
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rehabilitación avulsion
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Pelvic Floor Disorders; Ultrasound Therapy; Complications; Physical Disorder; Obstetric Labor Complications
MeSH Terms: conditions — Pelvic Floor Disorders; Obstetric Labor Complications

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The therapy lasted two months, at a rate of two sessions per week, with a duration of 45 minutes per session. The program consisted of pelvic floor exercises assisted by manometric biofeedback, which were performed in supine position for 20 minutes. In addition, active lumbopelvic stabilization exercises, including the contraction of pelvic floor muscles was performed in supine, plank and quadruped position.
  Together with the treatment at the clinic, patients were asked to perform a series of exercises at home, consisting in: 8-12 sustained contractions of 6 seconds, with a subsequent rest period of double the work-time, followed by 3-5 fast contractions of 2 seconds with maximum intensity, resting double the work-time. Domiciliary exercises were performed in supine, siting and standing position.
  Interventions: Other: Physiotherapy treatment
- Control group (No Intervention): The control group received an information brochure with recommendations, including the same program of pelvic floor exercises taught to the patients in the experimental group, but without carrying out any kind of supervision by the physiotherapist.

INTERVENTIONS:
Other: Physiotherapy treatment — Physiotherapy treatment consisted of pelvic floor exercises assisted by manometric biofeedback. In addition, active lumbopelvic stabilization exercises, including the contraction of pelvic floor muscles was performed in supine, plank and quadruped position.
  Arms: Experimental group

SUMMARY:
SUMMARY: (Objective, design, scope of the study, subjects of study, instrumentation, results, conclusions)

Objectives: To evaluate if the physiotherapy treatment in pelvic floor dysfunctions, identified by transperineal ultrasound 3 / 4D, in postpartum improve the tone and functionality of pelvic floor.

Design: Post-authorization, prospective, longitudinal randomized intervention study

Scope: Full-term deliveries at the University Hospital. Subjects of study: Full-term primiparous and full-term pregnancies with pelvic floor lesion, identified by transperineal ultrasound 3 / 4D, which are randomized between the physiotherapy treatment of pelvic floor and the non-work.

Variables: Primary variable: Assess the improvement in contractility / tone, evaluation by manometry and assess the anatomical improvement of the area of ?? the genital hiatus, stay by transperineal ultrasound 3 / 4D. Secondary variables: Identify the levator ani muscle injury rate, estimate the sonographic changes in the levator ani muscle through rehabilitation. Analyze the improvement of the symptoms associated with the public organic prolapse and evaluate the improvement of the quality of life.

Data analysis: To detect a difference of 10% in the reduction of the size of the index between the study groups (not intervened / intervened) after 6 months of intervention, standard deviation 10%, Error-alpha 5%, Error- beta 10% (P90%) we need 23 women in each group. Assuming a loss of 10% in the follow-up, the final size would be 52 women, 26 per group.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery
* Cephalic presentation
* Primiparity
* At term gestation (37-42 weeks)
* No prior pelvic floor corrective surgery
* Written informed consent

Exclusion Criteria:

* Pregnancies with severe maternal or fetal pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Contractility | 6 months after randomisation
  Assess the improvement in contractility / tone, evaluated by manometry, of the pelvic floor produced by the treatment of postpartum physiotherapy of the pelvic floor.

SECONDARY OUTCOMES:
Changes in the levator ani muscle | 6 months after randomisation
  To estimate the ultrasonographic changes in the levator ani muscle after rehabilitation, determining the maximum thicknesses and levator ani muscle area.

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio García Mejido, Principal Investigator — Hospital Universitario Nuestra Señora de Valme
Locations (1):
- Hospital Nuestra Señora de Valme, Seville, Spain